CLINICAL TRIAL: NCT05807828
Title: The Role of Virtual Reality Simulation in Acquiring Basic Surgical Skills in Total Hip Arthroplasty by Medical Students- a Prospective Randomized Clinical Trial
Brief Title: VR Simulation and Basic Skills in THA
Acronym: MD-VR-THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: ORamaVr SA ( Switzerland) (Unknown)
Responsible Party: Principal Investigator, Eustathios Kenanidis, Assistant Professor of Orthopaedic Surgery & Traumatology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 79/2023
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Educational Problems; Hip Arthroplasty; Osteoarthritis, Hip; Medical Students
Keywords: virtual reality; hip arthroplasty; surgical skills; medical students
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: All participants will be randomized to the VR simulation or control group for cup inclination and stem version assessment by a computerized random number generator. The VR group will perform implantation on sawbones after VR education and the control group without VR education.
Who Masked: Outcomes Assessor
Masking Description: The personnel that will assess the cup inclination and stem version will not know the group assignment of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): This group will include medical students who will only watch instructional videos on basic THA skills on the cup or stem implantation before actual implantation on sawbones
  Interventions: Procedure: VR simulation on basic THA skills
- VR Group (Other): This group will include medical students who will watch instructional videos and perform three consecutive VR sessions on basic THA skills on the cup or stem implantation before actual implantation on sawbones
  Interventions: Procedure: VR simulation on basic THA skills

INTERVENTIONS:
Procedure: VR simulation on basic THA skills — The medical students' VR group will perform three VR simulation sessions on basic THA skills on the cup or stem implantation before actual implantation.

SUMMARY:
This prospective randomised clinical trial aims to test if virtual reality (VR) simulation helps acquire basic surgical skills in total hip arthroplasty (THA) by medical students.

The main question[s] it aims to answer are:

1. Can VR simulation develop the medical students' basic surgical skills and medical knowledge in THA?
2. Will VR simulation become a part of orthopaedic surgical education?

Participants will be randomised into two groups (VR and control).

1. They will be asked to watch a very detailed video explaining basic rules and skills in implanting the acetabular cup and femoral stem in THA
2. The VR group will perform at least three VR THA sessions concerning cup (inclination) and stem (version) implantation
3. Then all participants will be asked to implant a cup and a stem in a predefined inclination and version, respectively, in sawbones
4. The mean difference between the predefined and the actual implanted cup inclination and version of the stem will be compared between groups

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial and received approval from the A.U.Th. Institutional Review Board.

Eligible study participants include undergraduate medical students at our university.

Exclusion criteria include a. postgraduate medical students b. prior experience in THA or general surgery.

One week before the planned VR-THA surgery session, all eligible A.U.Th. Medical students will be invited to an information session regarding the study and will be voluntarily enrolled, providing inform consent.

Medical students were explicitly chosen for participation because they are surgically naïve and would most likely benefit from basic skills training in THA.

Immediately after enrollment, medical students will be asked to complete a multiple-choice pretest to quantify their baseline medical and procedural knowledge of hip arthritis and THA. All participants will be unaware and unable to prepare for the pretest assessment, which allows the test scores to be considered an accurate measure of baseline knowledge.

The medical students will be asked to watch a detailed video explaining basic rules and skills for implanting the acetabular cup and femoral stem in THA. The video will be focused on practices and methods to achieve specific cup inclination and stem version during implantation.

All participants will be randomized to the VR simulation or control group for cup inclination assessment by a computerized random number generator. Participants will be privately notified of their randomization by e-mail and asked not to disclose their designated cohort with any other study participant or research personnel. Only a research team member will be aware of the cohort assignments during this study. The participants enrolled on the VR group for cup inclination will be the control group for the stem version group and vice versa.

Before the VR-THA, participants will be asked to complete a survey evaluating their previous video games and VR technology experience.

All control group participants will then be asked to implant a cup or a stem in a predefined inclination and version in sawbones. The cup inclination and stem version will be evaluated using specific goniometers and assessment of photographs taken during implantation. The evaluation will be performed by study personnel unaware of the participants' group assignment.

All VR group participants will then be asked to complete three consecutive VR sessions using the VR system (ORama VR, Geneva, Switzerland), performing cup or stem implantation based on their group. All VR group participants will then be asked to implant a cup or a stem in a predefined inclination and version in sawbones. The cup inclination and stem version will be evaluated using the same specific goniometers and assessment of photographs that will be taken during implantation. The evaluation will be performed by the same study personnel unaware of the participants' group assignment. This personnel will also record the time needed for implantation.

During implantation in sawbones, a study assistant will be present who will be instructed to intervene only if the study participants request assistance or cannot progress through the task.

Upon completion of the VR-THAs, participants will complete a survey focused on their interest in using VR simulations for surgical skills training and assessing for potential negative consequences. Power analysis was performed, indicating that more than 30 participants will be necessarily enrolled in each group.

The primary outcome will be the mean difference between the asked predefined and the actual implanted cup inclination or cup version between the control and VR groups.

The secondary outcomes will be

1. the percentage difference of the target approach between the asked and the actual implanted cup inclination or cup version for each participant performing implantation (one task will be performed as the VR and the other as the control group).
2. Differences in completing the task between groups will also be recorded ( time needed to complete the task and asking for assistance).

ELIGIBILITY:
Inclusion criteria:

a. undergraduate medical students at Aristotle University of Thessaloniki

Exclusion criteria:

1. postgraduate medical students
2. prior experience in THA or general surgery.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2023-03-26 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleftherios Tsiridis, Professor, Principal Investigator — Aristotle University Medical School
Locations (1):
- Aristotle University Medical School, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
The data will be available to other researchers upon publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon publication and forever
Access Criteria: Upon publication and forever

REFERENCES:
- [Background] Logishetty K, Rudran B, Cobb JP. Virtual reality training improves trainee performance in total hip arthroplasty: a randomized controlled trial. Bone Joint J. 2019 Dec;101-B(12):1585-1592. doi: 10.1302/0301-620X.101B12.BJJ-2019-0643.R1. PMID 31786991
- [Result] Hooper J, Tsiridis E, Feng JE, Schwarzkopf R, Waren D, Long WJ, Poultsides L, Macaulay W; NYU Virtual Reality Consortium. Virtual Reality Simulation Facilitates Resident Training in Total Hip Arthroplasty: A Randomized Controlled Trial. J Arthroplasty. 2019 Oct;34(10):2278-2283. doi: 10.1016/j.arth.2019.04.002. Epub 2019 Apr 8. PMID 31056442
- [Result] Logishetty K, Gofton WT, Rudran B, Beaule PE, Cobb JP. Fully Immersive Virtual Reality for Total Hip Arthroplasty: Objective Measurement of Skills and Transfer of Visuospatial Performance After a Competency-Based Simulation Curriculum. J Bone Joint Surg Am. 2020 Mar 18;102(6):e27. doi: 10.2106/JBJS.19.00629. PMID 31929324
- [Derived] Kenanidis E, Boutos P, Voulgaris G, Zgouridou A, Gkoura E, Gamie Z, Papagiannakis G, Tsiridis E. Effectiveness of virtual reality compared to video training on acetabular cup and femoral stem implantation accuracy in total hip arthroplasty among medical students: a randomised controlled trial. Int Orthop. 2024 Mar;48(3):625-633. doi: 10.1007/s00264-023-06038-8. Epub 2023 Nov 23. PMID 37993676

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group for Cup Training and VR Group for Stem Training: This group include medical students who only watched instructional videos on basic THA skills on the cup implantation before actual implantation on sawbones. These students also watched instructional videos and performed three consecutive VR sessions on basic THA skills on the stem implantation before actual implantation on sawbones.
- VR Group for Cup Training and Control Group for Stem Training: This group include medical students who watched instructional videos and perform three consecutive VR sessions on basic THA skills on the cup implantation before actual implantation on sawbones. These students also watched only instructional videos on basic THA skills on the stem implantation before actual implantation on sawbones.
Period: Overall Study
Arm/Group | Control Group for Cup Training and VR Group for Stem Training | VR Group for Cup Training and Control Group for Stem Training
Started | 54 | 47
Completed | 54 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group for Cup Training and VR Group for Stem Training | VR Group for Cup Training and Control Group for Stem Training | Total
Number analyzed (Participants) | 54 | 47 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.26 (2.896) | 23.49 (3.035) | 23.37 (2.949)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 32 | 24 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 54 | 47 | 101
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Greece | 54 | 47 | 101
Years of medical school attended [Count of Participants; unit: Participants] — Medical students were asked to complete a multiple-choice pretest determining their school age.
  Participants
    1 year of medical school attended | 2 | 3 | 5
    2 years of medical school attended | 5 | 4 | 9
    3 years of medical school attended | 7 | 4 | 11
    4 years of medical school attended | 12 | 13 | 25
    5 years of medical school attended | 24 | 19 | 43
    6 years of medical school attended | 4 | 4 | 8
Previous VR technology experience [Number; unit: participants]
  Previous participation in a vr training programme | 7 | 3 | 10
  Previous experience with vr headset | 28 | 16 | 44
  Owning a vr headset | 2 | 0 | 2
  Having general knowledge about vr technology | 53 | 47 | 100
Medical and procedural knowledge of hip arthritis and THA [Number; unit: participants]
  Previous attendance at orthopaedic surgery | 16 | 10 | 26
  Previous education on a surgical procedure (not orthopaedic) | 15 | 10 | 25
  Having knowledge of what a hip arthroplasty involves (femoral stem, femoral head, etc.) | 45 | 37 | 82
  Having knowledge of the pathophysiology of osteoarthritis | 42 | 38 | 80
  Having knowledge of the fixation materials for hip arthroplasty | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Medical Students Surgical Skills Differences Between VR and Control Group.
Description: The primary outcome will be the mean difference between the asked predefined and the actual implanted cup and stem inclination or version between the Control and VR groups.
  After completing VR training, all participants were asked to implant the cup at a 60-degree inclination in sawbones and the femoral stem at 20 degrees of anteversion. The cup inclination and stem version were evaluated using goniometers and performed by study personnel unaware of the participant's group assignment. To determine the cup inclination and femoral stem version angles, we utilised a hemipelvis and a femoral sawbone, clamps, an acetabular cup and a femoral rasp with an insertion handle, and a standard goniometer. So, the primary outcome was the mean difference between the asked predefined (60 degrees cup inclination/ 20 degrees stem anteversion) and the actual implanted cup and stem inclination or version by the students on sawbones between the Control and VR groups.
Time Frame: 2 Months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Group for Cup Training and VR Group for Stem Training | VR Group for Cup Training and Control Group for Stem Training
Number analyzed (Participants) | 54 | 47
degrees
  Cup Implantation (mean) | 51.5 (12.4) | 59.1 (6.1)
  Stem Implantation (mean) | 115.9 (142.8) | 201.5 (156.3)
Statistical Analysis 1: Comparison: Control Group for Cup Training and VR Group for Stem Training vs VR Group for Cup Training and Control Group for Stem Training; The median difference between the cup angle of the Control Group for Cup Training and the cup angle of VR Group for Cup Training; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 7.5
Statistical Analysis 2: Comparison: Control Group for Cup Training and VR Group for Stem Training vs VR Group for Cup Training and Control Group for Stem Training; The median difference between the stem angle of the Control Group for Stem Training and the stem angle of VR Group for Stem Training; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 291.5

2. Secondary Outcome: Surgical Skills Differences in Implantation Following VR Training vs. No Training
Description: This secondary outcome will assess the difference between the target and actual implantations performed by students with or without VR training. Each medical student performed two implantations, one with and the other without VR training. The implantation with VR training was assessed in the VR group and the other in the control group. All implantations following VR training were included in the VR group, and those without VR training were included in the Control group. For this measurement, the cup or stem implantation was not evaluated. Each group included both stem and cup implantations, based on whether VR was used or not for the implantation. We had just one value for each arm, rather than multiple assessments. We will report deviations from the predefined target of implantation, presenting the data individually in degrees of deviation.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- VR Group: This group include all medical students (47 of them performed cup implantation following VR training and 54 performed stem implantation following VR training).
- Control Group: This group include all medical students (47 of them performed stem implantation without VR training and 54 performed cup implantation without VR training).
Arm/Group | VR Group | Control Group
Number analyzed (Participants) | 101 | 101
degrees | 54.5 (106.6) | 89.8 (133.9)
Statistical Analysis 1: Comparison: VR Group vs Control Group; Each medical student carried out an implantation following VR training and without VR training. Therefore, there was a deviation (mean difference) between the predefined target and the implanted inclination for the cup or the stem version for the same medical student with VR training; Test type: Superiority; p < 0.05, paired t-test; Mean Difference (Final Values) = 54.5, Standard Deviation 106.6
Statistical Analysis 2: Comparison: VR Group vs Control Group; Each medical student carried out an implantation following VR training and without VR training. Therefore, there was a deviation (mean difference) between the predefined target and the implanted inclination for the cup or the stem version for the same medical student without VR training (control); Test type: Superiority; p < 0.05, paired t-test; Mean Difference (Final Values) = 89.8, Standard Deviation 133.9

3. Secondary Outcome: Time Needed to Perform Each Task
Description: Time needed for implantation from each participant was recorded both for stem and cup. Each participant performed one implantation following a previous VR training and another without training. Both times were recorded.
Time Frame: seconds
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control Group for Cup Training and VR Group for Stem Training | VR Group for Cup Training and Control Group for Stem Training
Number analyzed (Participants) | 54 | 47
seconds
  Time needed for cup implantation for Control cup and VR cup groups | 35 (27) | 21 (25)
  Time needed for stem implantation for VR stem and Control stem groups | 43 (46) | 45 (37)
Statistical Analysis 1: Comparison: Control Group for Cup Training and VR Group for Stem Training vs VR Group for Cup Training and Control Group for Stem Training; Median difference between the time needed for cup implantation for Control cup group and the time needed for cup implantation for VR cup group; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 14
Statistical Analysis 2: Comparison: Control Group for Cup Training and VR Group for Stem Training vs VR Group for Cup Training and Control Group for Stem Training; Median difference between the time needed for stem implantation for Control stem group and the time needed for stem implantation for VR stem group; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2

ADVERSE EVENTS:
Time Frame: The study takes 2 months to complete. Our study is a non-intervention study performed by medical students in sawbones, so no adverse event is expected.
Description: Our study did not include any intervention for the participants. All students simply watch training videos or conduct VR sessions and then test their knowledge on sawbones. Our study is a non-intervention study performed by medical students in sawbones, so no adverse event is expected. So it makes sense that there are no adverse effects at all in our study. There is no mortality or other adverse event risk. This is the reason that 0% of the students are risk of adverse events.
Arm/Group | Control Group for Cup Training and VR Group for Stem Training | VR Group for Cup Training and Control Group for Stem Training
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/47
Other Adverse Events (participants affected / at risk) | 0/54 | 0/47

LIMITATIONS AND CAVEATS:
Limitations

1. We used medical students and not junior resident surgeons which may be more appropriate for this study. Medical students are completely naïve to these procedures, more easily found and not subjected to surgical operations. This controlled environment will not be available during residency.
2. The Saw Bone model and the VR environment are not completely accurate representations of an actual surgical scenario.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT05807828/Prot_SAP_000.pdf